CLINICAL TRIAL: NCT02288065
Title: Predictive Factors and Outcome in Medical Thoracoscopy
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Yserbyt Jonas, MD, KU Leuven
Other Study IDs: S561430
Record Dates: First submitted 2014-11-04; First posted 2014-11-11 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Pleuritis
MeSH Terms: conditions — Pleurisy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- responders: amelioration of dyspnea radiological amelioration after sterile talc pleurodesis
  Interventions: Drug: sterile talc pleurodesis
- failed intervention: unchanged symptoms and radiology after sterile talc pleurodesis
  Interventions: Drug: sterile talc pleurodesis

INTERVENTIONS:
Drug: sterile talc pleurodesis — medical thoracoscopy and talc pleurodesis. No specific device is studied.
  Other Names: medical thoracoscopy

SUMMARY:
Retrospective survey for factors predicting the outcome of medical thoracoscopy

DETAILED DESCRIPTION:
Retrospective survey for factors predicting the outcome of medical thoracoscopy in patients with malignant pleuritis

ELIGIBILITY:
Inclusion Criteria:

* progressive malignancy
* pleuritis

Exclusion Criteria:

* respiratory failure
* unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pulmonary or extrathoracic malignancy
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Chest X-ray | 3 months
  radiological resolution of pleuritis; 3 level severity grading (A, B, C, with C as worst grade)

SECONDARY OUTCOMES:
time interval | 12 months
  survival in months

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Yserbyt, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium